CLINICAL TRIAL: NCT00464984
Title: Lifestyle Intervention in Morbidly Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital of Vestfold (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Jøran Hjelmesæth, Head of Morbid Obesity Centre, The Hospital of Vestfold
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-05175.1
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Morbid Obesity
Keywords: Weight loss; Physical fitness; Quality of life
MeSH Terms: conditions — Obesity, Morbid; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ILI-group (Active Comparator): Intensive lifestyle intervention at a tertiary care rehabilitation center. Treatment included changes in both dietary habits (calori restriction) and physical activity with particularly high intensity the first 3 months.
  Interventions: Behavioral: Lifestyle intervention
- MLI (Active Comparator): Moderate lifestyle intervention at a secondary care outpatient center. Treatment included moderate changes in dietary habits (calori restriction) and physical activity.
  Interventions: Behavioral: Lifestyle intervention

INTERVENTIONS:
Behavioral: Lifestyle intervention — Intensive lifestyle intervention at a rehabilitation centre 3 times a week the first 3 months of study

SUMMARY:
The long term effects of organized lifestyle intervention on weight loss, physical fitness and quality of life in morbidly obese patients have not been extensively studied. The objective of this study is to investigate whether an intensive lifestyle intervention program in a tertiary care clinic (Spesialsykehuset for Rehabilitating) is superior to lifestyle intervention in a primary care setting with respect to long term (4-years) changes in weight loss, physical fitness and quality of life

DETAILED DESCRIPTION:
Due to limited recruitment from GP, the study design has been changed into an observational long term study following the participants in the intensive lifestyle intervention group

ELIGIBILITY:
Inclusion Criteria:

* Morbidly obese patients not planned for bariatric surgery

Exclusion Criteria:

* Participation in other weight loss programs during the last 12 mths
* Serious psychiatric conditions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-08; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Weight loss, physical fitness and quality of life | 1 and 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Jøran Hjelmesæth, MD, PhD, Study Chair — Morbid Obesity Center, Hospital of Vestfold, Boks 2168, NORWAY
Locations (1):
- Spesialsykehuset for Rehabilitering i Stavern, Stavern, Vestfold, Norway